CLINICAL TRIAL: NCT06701695
Title: Efficacy of Intraoperative Periarticular Injections in Reducing Blood Loss and Transfusion Requirements in Hip Fracture Hemiarthroplasty: A Randomized Controlled Trial
Brief Title: Efficacy of Intraoperative Periarticular Injections in Hip Fracture Hemiarthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, TANER KARLIDAĞ, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-ORT-TK-01
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Femoral Neck Fractures; Hemiarthroplasty; Blood Loss Requiring Transfusion
Keywords: Hip Fracture; Hemiarthroplasty; Periarticular injection; Blood loss; Blood transfusion requirement
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Two groups were established, one serving as the control group receiving standard hemiarthroplasty treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the trial, patients were kept unaware of their group assignments, ensuring they remained blinded to the study parameters. While the surgeon possessed knowledge of the group allocations, he was not directly involved in patient data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periarticular injection group (Active Comparator): Patients in the periarticular injection group were administered a 100 mL periarticular solution comprising 200 mg of bupivacaine (40 mL), 60 mg of ketorolac (2 mL), 8 mg of dexamethasone (2 mL), 2 mg of 1:1000 epinephrine (2 mL), and standard saline solution (54 mL). This solution was prepared in two 50 mL syringes. The first syringe containing 50 mL of the cocktail was injected into the capsule and gluteal muscles before femoral stem insertion. Following joint capsule closure, the second syringe containing 50 mL of the periarticular injection cocktail was infiltrated into the fascia lata muscle, subcutaneous tissue, and wound layers.
  Interventions: Procedure: Periarticular Injection (PAI); Procedure: Control (Standard treatment)
- Control group (Sham Comparator): Participants in the control group underwent standard hemiarthroplasty treatment, with no administration of periarticular injections.
  Interventions: Procedure: Control (Standard treatment)

INTERVENTIONS:
Procedure: Periarticular Injection (PAI) — Patients in the periarticular injection group were administered a 100 mL periarticular solution comprising 200 mg of bupivacaine (40 mL), 60 mg of ketorolac (2 mL), 8 mg of dexamethasone (2 mL), 2 mg of 1:1000 epinephrine (2 mL), and standard saline solution (54 mL). This solution was prepared in two 50 mL syringes. The first syringe containing 50 mL of the cocktail was injected into the capsule and gluteal muscles prior to femoral stem insertion. Following joint capsule closure, the second syringe containing 50 mL of the periarticular injection cocktail was infiltrated into the fascia lata muscle, subcutaneous tissue, and wound layers.
  Arms: Periarticular injection group
Procedure: Control (Standard treatment) — The control group received the conventional treatment protocol.

SUMMARY:
The objective of this study was to assess the effectiveness of the intraoperative periarticular solution in reducing blood loss and minimizing transfusion requirements in patients with femoral neck fractures who underwent hemiarthroplasty.

DETAILED DESCRIPTION:
Hip fractures in the elderly represent a significant public health challenge, marked by elevated rates of morbidity and mortality. The worldwide increase in life expectancy has led to a corresponding rise in the incidence of hip fractures. Notably, increased perioperative blood loss has been identified as a critical factor that heightens the risk of complications and mortality. Consequently, contemporary research efforts have focused on addressing this pivotal issue. Various strategies have been developed, including controlled hypotensive anesthesia and the utilization of pharmacological agents aimed at reducing the perioperative blood products. The necessity for the efficacy of tranexamic acid (TXA) in mitigating blood loss has been well-established across numerous surgical specialties. This study is motivated by the need for an effective and safe approach to perioperative blood salvage. To date, there appears to be a lack of research examining the effectiveness of the intraoperative periarticular injection technique (100 mL periarticular solution comprising 200 mg of bupivacaine (40 mL), 60 mg of ketorolac (2 mL), 8 mg of dexamethasone (2 mL), 2 mg of 1:1000 epinephrine (2 mL), and standard saline solution (54 mL). This solution was prepared in two 50 mL syringes. The first syringe containing 50 mL of the cocktail was injected into the capsule and gluteal muscles before femoral stem insertion. Following joint capsule closure, the second syringe containing 50 mL of the periarticular injection cocktail was infiltrated into the fascia lata muscle, subcutaneous tissue, and wound layers) regarding blood loss reduction. Therefore, this study aims to investigate the following questions: 1) Is intraoperative periarticular injection an effective technique for minimizing blood loss in patients with hip fractures? and 2) What proportion of the salvaged blood loss can be attributed to hidden blood loss?

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of femoral neck fracture

Exclusion Criteria:

* Anti-aggregant, anti-coagulant or anti-thrombotic therapy
* Pathological fractures, periprosthetic fractures, or revision procedures
* Intolerance or allergy to the medications utilized in the study
* Refused to participation

Ages: 58 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss | Preoperative and postoperative hematocrit (HCT) and hemoglobin (Hb) levels measured over the first three days
  The calculation of Total Blood Volume (TBV) was conducted using the following manner:
  TBV= k1 x H3 + k2 x W+ k3 For males, k1 = 0.3669, k2 = 0.03219, and k3 = 0.1833; for females, k1 = 0.3561, k2 = 0.03308, and k3 = 0.1833; H=height (m) and W=weight (kg)
  The calculation of Total blood loss (TBL) was conducted using the Gross formula method as follows:
  TBL= TBV x (Preoperative HCT (Hematocrit) - Postoperative 3-day HCT) / Mean HCT

SECONDARY OUTCOMES:
Hidden Blood Loss | Postoperative first three days
  Intraoperative Blood Loss (IBL) was determined through anesthesia recordings during the operation, which included measuring blood suction bottles and the weight of surgical swabs.
  Visible Blood Loss = Intraoperative Blood Loss + Postoperative suction drain volume The Total Hidden Blood Loss (HBL) volume was determined by deducting the visible blood loss volume from the TBL volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In the event that reviewers make such a request, participant data may be made available for sharing in the future.

REFERENCES:
- [Result] Keating EM. Preoperative evaluation and methods to reduce blood use in orthopedic surgery. Anesthesiol Clin North Am. 2005 Jun;23(2):305-13, vi-vii. doi: 10.1016/j.atc.2005.02.006. PMID 15922902
- [Result] Desai SJ, Wood KS, Marsh J, Bryant D, Abdo H, Lawendy AR, Sanders DW. Factors affecting transfusion requirement after hip fracture: can we reduce the need for blood? Can J Surg. 2014 Oct;57(5):342-8. doi: 10.1503/cjs.030413. PMID 25265109
- [Result] Liodakis E, Antoniou J, Zukor DJ, Huk OL, Epure LM, Bergeron SG. Major Complications and Transfusion Rates After Hemiarthroplasty and Total Hip Arthroplasty for Femoral Neck Fractures. J Arthroplasty. 2016 Sep;31(9):2008-12. doi: 10.1016/j.arth.2016.02.019. Epub 2016 Feb 17. PMID 26975602
- [Result] Moran CG, Wenn RT, Sikand M, Taylor AM. Early mortality after hip fracture: is delay before surgery important? J Bone Joint Surg Am. 2005 Mar;87(3):483-9. doi: 10.2106/JBJS.D.01796. PMID 15741611
- [Result] Carson JL, Poses RM, Spence RK, Bonavita G. Severity of anaemia and operative mortality and morbidity. Lancet. 1988 Apr 2;1(8588):727-9. doi: 10.1016/s0140-6736(88)91536-x. PMID 2895260
- [Result] Veronese N, Maggi S. Epidemiology and social costs of hip fracture. Injury. 2018 Aug;49(8):1458-1460. doi: 10.1016/j.injury.2018.04.015. Epub 2018 Apr 20. PMID 29699731
- [Result] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Result] Turan S, Bingol O. Is tranexamic acid effective on hidden blood loss in patients during total knee arthroplasty? Jt Dis Relat Surg. 2020;31(3):488-493. doi: 10.5606/ehc.2020.78024. PMID 32962580
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Result] Liu W, Deng S, Liang J. Tranexamic acid usage in hip fracture surgery: a meta-analysis and meta-regression analysis of current practice. Arch Orthop Trauma Surg. 2022 Oct;142(10):2769-2789. doi: 10.1007/s00402-021-04231-1. Epub 2021 Oct 28. PMID 34709457
- [Result] Li ZJ, Zhao MW, Zeng L. Additional Dose of Intravenous Tranexamic Acid after Primary Total Knee Arthroplasty Further Reduces Hidden Blood Loss. Chin Med J (Engl). 2018 Mar 20;131(6):638-642. doi: 10.4103/0366-6999.226884. PMID 29521284
- [Result] Smith GH, Tsang J, Molyneux SG, White TO. The hidden blood loss after hip fracture. Injury. 2011 Feb;42(2):133-5. doi: 10.1016/j.injury.2010.02.015. Epub 2010 Mar 16. PMID 20236640
- [Result] Watts CD, Houdek MT, Sems SA, Cross WW, Pagnano MW. Tranexamic Acid Safely Reduced Blood Loss in Hemi- and Total Hip Arthroplasty for Acute Femoral Neck Fracture: A Randomized Clinical Trial. J Orthop Trauma. 2017 Jul;31(7):345-351. doi: 10.1097/BOT.0000000000000837. PMID 28633147
- [Result] Baskaran D, Rahman S, Salmasi Y, Froghi S, Berber O, George M. Effect of tranexamic acid use on blood loss and thromboembolic risk in hip fracture surgery: systematic review and meta-analysis. Hip Int. 2018 Jan;28(1):3-10. doi: 10.5301/hipint.5000556. PMID 28983887
- [Result] Foss NB, Kehlet H. Hidden blood loss after surgery for hip fracture. J Bone Joint Surg Br. 2006 Aug;88(8):1053-9. doi: 10.1302/0301-620X.88B8.17534. PMID 16877605
- [Result] Ashkenazi I, Schermann H, Gold A, Lin R, Pardo I, Steinberg E, Sternheim A, Snir N. Tranexamic acid in hip hemiarthroplasty. Injury. 2020 Nov;51(11):2658-2662. doi: 10.1016/j.injury.2020.07.061. Epub 2020 Aug 1. PMID 32763019
- [Result] Amin NH, Hutchinson HL, Sanzone AG. Infiltration Techniques for Local Infiltration Analgesia With Liposomal Bupivacaine in Extracapsular and Intracapsular Hip Fracture Surgery: Expert Panel Opinion. J Orthop Trauma. 2018 Aug;32 Suppl 2:S5-S10. doi: 10.1097/BOT.0000000000001227. PMID 30028758
- [Result] Bentler SE, Liu L, Obrizan M, Cook EA, Wright KB, Geweke JF, Chrischilles EA, Pavlik CE, Wallace RB, Ohsfeldt RL, Jones MP, Rosenthal GE, Wolinsky FD. The aftermath of hip fracture: discharge placement, functional status change, and mortality. Am J Epidemiol. 2009 Nov 15;170(10):1290-9. doi: 10.1093/aje/kwp266. Epub 2009 Oct 4. PMID 19808632
- [Result] Li J, Dai F, Chang D, Harmon E, Ibe I, Sukumar N, Halaszynski TM, Rubin LE, O'Connor MI. A Practical Analgesia Approach to Fragility Hip Fracture: A Single-Center, Retrospective, Cohort Study on Femoral Nerve Block. J Orthop Trauma. 2019 Apr;33(4):175-179. doi: 10.1097/BOT.0000000000001391. PMID 30570615